CLINICAL TRIAL: NCT00405899
Title: Pilot Study of Allergy Immunotherapy and Prevention of Viral Respiratory Infections
Status: Completed | Type: Observational
Sponsor: West Penn Allegheny Health System (Other)
Collaborators: Pennsylvania Allergy and Asthma Research Foundation (Unknown)
Responsible Party: Deborah Gentile/Principal Investigator, Allegheny General Hospital
Other Study IDs: RC - 4064
Record Dates: First submitted 2006-11-28; First posted 2006-11-30 (Estimated); Last update posted 2010-05-31 (Estimated); Status verified 2010-05

CONDITIONS: Allergy; Seasonal Allergic Rhinitis; Perennial Allergic Rhinitis
Keywords: Allergy; Seasonal Allergic Rhinitis; Perennial Allergic Rhinitis
MeSH Terms: conditions — Hypersensitivity; Rhinitis, Allergic, Seasonal; Rhinitis, Allergic, Perennial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Immunotherapy: Patients starting immunotherapy
- Non-immunotherapy: Patients being treated using methods other than immunotherapy

SUMMARY:
The objective of this study is to determine whether there is a relationship between interferon-gamma levels and the incidence of viral respiratory infections in allergic children treated with allergy immunotherapy as compared to those treated with standard medical care (nasal steroids, antihistamines) over a 1-year period. The hypotheses to be tested are 1) interferon-gamma levels will be significantly increased 3, 6, 9 and 12 months in allergic children treated with allergy immunotherapy as compared to those treated with standard medical care, 2) the incidence of viral respiratory infections will be reduced at 3, 6, 9 and 12 months in allergic children treated with allergy immunotherapy as compared to those treated with standard medical care.

DETAILED DESCRIPTION:
This study will consist of five visits. Visit 1 will occur after subjects complete an initial clinical evaluation for allergy at this site. Subjects will select their treatment (allergy immunotherapy as compared to standard medical care) prior to enrollment in this study.

Visit 1 will include informed consent, review of inclusion and exclusion criteria and phlebotomy for the determination of serum interferon-gamma levels. At the end of this visit, diary cards to capture the frequency of symptoms of viral respiratory infections will be distributed. Visits 2-5 will occur 3, 6, 9 and 12 months after visit 1 and will include review/exchange of diary cards, and phlebotomy for determination of serial serum interferon-gamma levels.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-18 years of age
* History of allergic rhinitis as confirmed by previous allergy skin testing conducted within the past year
* Subjects assigned to the allergy immunotherapy must be prescribed therapy according to national recommendations using FDA-approved allergy extracts supplied by Greer Laboratories

Exclusion Criteria:

* Concurrent difficult to control asthma or an underlying immune deficiency

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Male and Female patients aged 6 to 18 years being treated for allergies.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2006-10; Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Gentile, MD, Principal Investigator — West Penn Allegheny Health System
Locations (1):
- Allegheny General Hospital, Pittsburgh, Pennsylvania, United States